CLINICAL TRIAL: NCT03724448
Title: Evaluation of the Efficacy of a Herbal Supplement in the Prevention of Treatment of Post-traumatic Stress Disorder Versus Placebo (PHYTéS Study)
Brief Title: The Efficacy of a Herbal Supplement in the Prevention of PTSD
Acronym: PHYTéS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hôpital Universitaire Sahloul (Other)
Responsible Party: Principal Investigator, Riadh Boukef, Professor, Hôpital Universitaire Sahloul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PHYTéS
Record Dates: First submitted 2018-06-24; First posted 2018-10-30 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: PTSD, Post Traumatic Stress Disorder; Diagnosis, Psychiatric; Follow up
MeSH Terms: conditions — Combat Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALEOZEN group (Experimental): Clinical information will be collected on a standardized card specifying general data on the patient, his antecedents, his telephone number, the circumstances of the traumatic event and the score of PDI, PDEQ and L-CROCQ, score PCL-5 to 10 days, 1 month and 6 months.
  Interventions: Drug: aleozen
- placebo group (Placebo Comparator): Clinical information will be collected on a standardized card specifying general data on the patient, his antecedents, his telephone number, the circumstances of the traumatic event and the score of PDI, PDEQ and L-CROCQ, score PCL-5 to 10 days, 1 month and 6 months.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: aleozen — treatment with herbal medicine
  Arms: ALEOZEN group
Drug: Placebo Oral Tablet — No aleozen treatment
  Arms: placebo group

SUMMARY:
Psycho-traumatic disorders are a disabling condition whose epidemiological data vary according to the country but also the populations studied and the measuring instruments used. The estimated prevalence of posttraumatic stress disorder (PTSD) appeared to be increasing in recent years, and this appears to be due, among other things, to the improvement of the standardized evaluation procedure. The survey "Mental Health in General Population", conducted in metropolitan France between 1999 and 2003 on more than 36,000 people estimated its instantaneous prevalence (last month) of a full PTSD was 0.7% in the SMPG overall sample, with almost equal frequency between men (45%) and women (55%). This figure is close to that reported in a European population for the ESEMeD study. A very significant psychiatric comorbidity was found in subjects with PTSD, particularly with mood disorders, other anxiety disorders and addictive behaviors. The link with the suicidal risk was clearly established, which is the gravity of this pathology.

The most important publications are made by American teams who have identified and evaluated the treatment of this pathology among veterans of the various wars led by the country.

DETAILED DESCRIPTION:
Psycho-traumatic disorders are a disabling condition whose epidemiological data vary according to the country but also the populations studied and the measuring instruments used. The estimated prevalence of posttraumatic stress disorder (PTSD) appeared to be increasing in recent years, and this appears to be due, among other things, to the improvement of the standardized evaluation procedure. The survey "Mental Health in General Population", conducted in metropolitan France between 1999 and 2003 on more than 36,000 people estimated its instantaneous prevalence (last month) of a full PTSD was 0.7% in the SMPG overall sample, with almost equal frequency between men (45%) and women (55%). This figure is close to that reported in a European population for the ESEMeD study. A very significant psychiatric comorbidity was found in subjects with PTSD, particularly with mood disorders, other anxiety disorders and addictive behaviors. The link with the suicidal risk was clearly established, which is the gravity of this pathology.

The most important publications are made by American teams who have identified and evaluated the treatment of this pathology among veterans of the various wars led by the country.

Barrois defines traumatic neurosis as "a group of psychological disorders that arise after a longer or shorter latency, following a very intense emotional shock".

Post-traumatic stress disorder is defined by the ICD-10 classification as a "delayed or prolonged" response to a stressful situation or event (short or long-term) that would provoke distress symptoms in anyone .

According to the American classification of the DSM-V, the diagnosis of PTSD is strictly established according to different criteria. Exposure to a traumatic event ("the person has been exposed, witnessed or confronted with an event or events that have involved death or death, or serious injury or threat to their physical integrity or 'others'), and reacting to it with a feeling of intense fear, helplessness or horror (criterion A). The event is constantly relived, manifested by at least one symptom of the repetition syndrome (criterion B) that can be repetitive and invasive memories of the event (including images, thoughts, perceptions), repetitive and painful dreams of the event, the impression or sudden acts "as if" the traumatic event recurred, an intense psychological distress when exposed to internal or external stimuli resembling an aspect of the trauma, a physiological reactivity during exposure to internal or external stimuli resembling or symbolizing an aspect of the trauma. Criterion C requires persistent avoidance of stimuli associated with trauma and blunting of general responsiveness (not present before trauma).

Criterion D refers to the impairment of cognition and mood associated with one or more traumatic events manifested by at least two symptoms, including dissociative amnesia, persistent and exaggerated negative self-perceptions of others, and world, a clear reduction of interest in important activities, a feeling of detachment and a persistent inability to feel positive emotions. There are also symptoms of neurovegetative activation, with at least two symptoms (criterion E) among sleep difficulties, irritability or anger, difficulty concentrating, hyper vigilance, startled reactions exaggerated. Criterion F concerns the duration of symptoms B, C and D which must exceed one month. The problem results in clinically significant distress or dysfunction at the social, occupational or other important operational level (criterion G). Criterion H eliminates that these symptoms are not due to the consumption of a substance (drug or alcohol) or another condition.

Despite this awareness of the functional impact of these psycho traumatic disorders, this pathology has remained under-identified both by health professionals and the general public and subsequently insufficiently treated, particularly in Tunisia. Several therapeutic protocols are proposed. The share of antidepressant treatments (yet first-line treatment in all international guidelines) is only 30% and the remaining 70% includes anxiolytics, hypnotics and herbal medicine. Several meta-analyzes have evaluated the efficacy of different families of antidepressants, but scientific research remains very poor in the field of herbal medicine.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who has been exposed to a traumatic event that could cause an acute PTSD (accident or aggression that causes intense fear, helplessness or horror)
* a PDI (Peri-traumatic Distress Inventory) score and / or PDEQ (Traumatic Traumatic Dissociation Experience Questionnaire - Evaluative Form)
* and / or (Appendix 1, 2 and 3) calculated between J1 and J3 and estimated moderate or high with a score> 15.

Exclusion Criteria:

* Any serious traumatized patient who needed treatment in intensive care.
* Any patient with psychiatric illness or psychotropic medication prior to randomization.
* Non-cooperating patient (unable to answer the assessment test).
* Non consenting patient.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
50% diminution or stabilization of CAPS score after 3 and 6 months | after 3 and 6 months of patient's inclusion
  50% diminution or stabilization of CAPS score

CONTACTS AND LOCATIONS:
Locations (1):
- HU Sahloul, sousse, Tunisia, Sousse, Itinéraire Ceinture Cité Sahloul, Tunisia

IPD SHARING:
Plan to Share IPD: No
researchers will participate in the recruitment of patients with post traumatic syndrom

REFERENCES:
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for prevention of post-traumatic stress disorder (PTSD) in individuals experiencing acute traumatic stress symptoms. Cochrane Database Syst Rev. 2024 May 20;5(5):CD013613. doi: 10.1002/14651858.CD013613.pub2. PMID 38767196
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for universal prevention of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2022 Feb 10;2(2):CD013443. doi: 10.1002/14651858.CD013443.pub2. PMID 35141873